CLINICAL TRIAL: NCT05549076
Title: Complicated Intra-abdominal Infections - the Greek Reality: a Prospective Observational Study
Brief Title: Hellenic Registry for cIAIs (HERCO-II)
Acronym: HERCO-II
Status: Completed | Type: Observational
Sponsor: Maximos Frountzas (Other)
Responsible Party: Sponsor-Investigator, Maximos Frountzas, Dr Maximos Frountzas MD MPA PhD, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Other Study IDs: HERCO-II 2022
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Intra-abdominal Infection
Keywords: complicated; intra-abdominal; infection; greek
MeSH Terms: conditions — Intraabdominal Infections; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complicated Intra-Abdominal Infections (cIAIs) represent an emergent surgical situation which lead to important non trauma-related mortality in several Emergency Surgical Centers worldwide. Their prevalence seemed to be unrelated to age, gender, health status and socioeconomic condition. Early diagnosis, timely septic source control, wide-spectrum antibiotic delivery and resuscitation with fluids and vasoactive agents in critically ill patients are fundamentals for successful cIAIs management. Moreover, septic shock, antibiotic resistant multi-pathogens and comorbidities have been associated with increased morbidity and mortality of cIAIs.

Several international health associations announce updated guidelines for cIAIs management. Nevertheless, such guidelines could not be widely implemented, because of specific features of several healthcare systems worldwide. The aim of the present study is to investigate the prevalence of cIAIs among the Greek health system and the potential association of time interval of septic source control, preoperative resuscitation and multidrug resistant pathogens with morbidity, mortality, ICU stay and length of stay in patients with cIAIs.

DETAILED DESCRIPTION:
Registry of patients with complicated intra-abdominal infections including:

* Patient demographics (gender, age, Carlson Comorbidity Index, cancer history/chemotherapy during the last 6 months, health unit stay during the last 6 months)
* Management (conservative, minimally invasive, surgical)
* Minimally invasive procedure - type (CT-guided drainage, endoscopic)
* Surgical procedure - type (open or laparoscopic, day or night, procedure description)
* Cultures (blood, peritoneal fluid, tissue)
* Time of diagnosis (respiratory rate, heart rate, systolic blood pressure, lactate acid in blood gases, temperature, white cell count, CRP)
* Just before procedure (respiratory rate, heart rate, systolic blood pressure, lactate acid in blood gases, vasoactive agent delivery, intubation)
* Intraoperative parameters (time interval between diagnosis and intervention, WSES score, operative time, open abdomen, VAC)
* After procedure (respiratory rate, heart rate, systolic blood pressure, lactate acid in blood gases, temperature, vasoactive agent delivery, intubation)
* Empirical wide-spectrum antibiotics (type and time interval from diagnosis)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Signed consent from patient or authorized representative
3. Complicated Intra-Abdominal Infection

   * Acute appendicitis with localized or diffuse peritonitis
   * Grade II or Grade III acute cholecystitis (Tokyo guidelines)
   * Visceral organ perforation with peritonitis
   * Bowel perforation after colonoscopy
   * Complicated diverticulitis (WSES classification)
   * Anastomotic leaks with abscess, localized or diffuse peritonitis

Exclusion Criteria:

1. Age < 18 years old
2. No signed consent from patient or authorized representative

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with complicated intra-abdominal infections.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Morbidity | 30 days
  Overall complications due to complicated intra-abdominal infections

SECONDARY OUTCOMES:
Mortality | 30 days
  Number of deaths due to complicated intra-abdominal infections
Length of stay | 30 days
  Days of hospitalization
Length of ICU stay | 30 days
  Days in the ICU
Organ failure | 30 days
  Dysfunction of one ore more organs
Re-operation rate | 30 days
  Re-operations after first surgical procedure
Multidrug resistant pathogen cultures | 30 days
  Results of pathogen cultures indicating multi-drug resistant variants.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos G Toutouzas, MD PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Hippocration General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shrestha B, Dunn L. The Declaration of Helsinki on Medical Research involving Human Subjects: A Review of Seventh Revision. J Nepal Health Res Counc. 2020 Jan 21;17(4):548-552. doi: 10.33314/jnhrc.v17i4.1042. PMID 32001865
- [Background] Ahmed S, Wilcox MH, Kirby A. Measuring outcomes in complicated intra-abdominal infections. Curr Opin Gastroenterol. 2020 Jan;36(1):1-4. doi: 10.1097/MOG.0000000000000591. PMID 31567430
- [Background] Leone S, Damiani G, Pezone I, Kelly ME, Cascella M, Alfieri A, Pace MC, Fiore M. New antimicrobial options for the management of complicated intra-abdominal infections. Eur J Clin Microbiol Infect Dis. 2019 May;38(5):819-827. doi: 10.1007/s10096-019-03533-y. Epub 2019 Mar 23. PMID 30903538
- [Background] Mayumi T, Okamoto K, Takada T, Strasberg SM, Solomkin JS, Schlossberg D, Pitt HA, Yoshida M, Gomi H, Miura F, Garden OJ, Kiriyama S, Yokoe M, Endo I, Asbun HJ, Iwashita Y, Hibi T, Umezawa A, Suzuki K, Itoi T, Hata J, Han HS, Hwang TL, Dervenis C, Asai K, Mori Y, Huang WS, Belli G, Mukai S, Jagannath P, Cherqui D, Kozaka K, Baron TH, de Santibanes E, Higuchi R, Wada K, Gouma DJ, Deziel DJ, Liau KH, Wakabayashi G, Padbury R, Jonas E, Supe AN, Singh H, Gabata T, Chan ACW, Lau WY, Fan ST, Chen MF, Ker CG, Yoon YS, Choi IS, Kim MH, Yoon DS, Kitano S, Inomata M, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: management bundles for acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):96-100. doi: 10.1002/jhbp.519. Epub 2017 Dec 16. PMID 29090868
- [Background] Sartelli M, Weber DG, Kluger Y, Ansaloni L, Coccolini F, Abu-Zidan F, Augustin G, Ben-Ishay O, Biffl WL, Bouliaris K, Catena R, Ceresoli M, Chiara O, Chiarugi M, Coimbra R, Cortese F, Cui Y, Damaskos D, De' Angelis GL, Delibegovic S, Demetrashvili Z, De Simone B, Di Marzo F, Di Saverio S, Duane TM, Faro MP, Fraga GP, Gkiokas G, Gomes CA, Hardcastle TC, Hecker A, Karamarkovic A, Kashuk J, Khokha V, Kirkpatrick AW, Kok KYY, Inaba K, Isik A, Labricciosa FM, Latifi R, Leppaniemi A, Litvin A, Mazuski JE, Maier RV, Marwah S, McFarlane M, Moore EE, Moore FA, Negoi I, Pagani L, Rasa K, Rubio-Perez I, Sakakushev B, Sato N, Sganga G, Siquini W, Tarasconi A, Tolonen M, Ulrych J, Zachariah SK, Catena F. 2020 update of the WSES guidelines for the management of acute colonic diverticulitis in the emergency setting. World J Emerg Surg. 2020 May 7;15(1):32. doi: 10.1186/s13017-020-00313-4. PMID 32381121